CLINICAL TRIAL: NCT06197971
Title: Comparative Effects of Instrument Assisted Soft Tissue Mobilization and Therapeutic Cupping on Hamstring Tightness Among Football Players
Brief Title: Instrument Assisted Soft Tissue Mobilization vs Therapeutic Cupping on Hamstring Tightness Among Football Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0461
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Flexibility; Hamstring Tightness; Instrument Assisted Soft Tissue Mobilization; Range of Motion
Keywords: Flexibility; Hamstring Tightness; Instrument Assisted Soft Tissue Mobilization; Cupping Technique; Football Players

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trail
Who Masked: Outcomes Assessor
Masking Description: The assessor who will take the readings is blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instrument Assisted Soft Tissue Mobilization (Other): The therapist will assess the hamstrings to identify areas of restriction or dysfunction. They will use the Graston Technique instruments to apply strokes and movements along the length of the muscle fibers. Sweeping strokes, cross-fiber friction, and circular motions patterns will be applied. The duration of the IASTM treatment will be 15-30 minutes.
  Interventions: Other: Instrument Assisted Soft Tissue Mobilization
- Therapeutic Cupping Technique (Other): After thorough assessment of the Hamstring area, a thin layer of lubricant will be applied on the area about to be cupped. Stationary cupping technique will be used for a duration of 5-15 minutes with multiple Silicone Cups applied on the Hamstrings. For cupping the hamstrings, cups with a diameter of around 1.5 to 2.5 inches (3.8 to 6.4 cm) will be suitable considering the large area of treatment
  Interventions: Other: Therapeutic Cupping Technique

INTERVENTIONS:
Other: Instrument Assisted Soft Tissue Mobilization — Graston Technique instruments to apply strokes and movements along the length of the muscle fibers. Sweeping strokes, cross-fiber friction, and circular motions patterns will be applied on hamstring muscles.
  Arms: Instrument Assisted Soft Tissue Mobilization
Other: Therapeutic Cupping Technique — Stationary cupping technique will be used for a duration of 5-15 minutes with multiple Silicone Cups applied on the Hamstrings.
  Arms: Therapeutic Cupping Technique

SUMMARY:
The study is randomized and single-blinded. Ethical approval is taken from ethical committee of Riphah International University, Lahore. Participants who meet the inclusion criteria will be enrolled and allocated in group A & B through sealed envelope method by Non-probability Convenient random sampling technique. Subjects in Group A will receive Instrument Assisted Soft Tissue Mobilization. Group B will receive Therapeutic Cupping.

DETAILED DESCRIPTION:
The objective of the study is to determine the effects of Instrument Assisted Soft Tissue Mobilization and Therapeutic Cupping on Hamstring tightness among football players. The study is randomized and single-blinded. Ethical approval is taken from ethical committee of Riphah International University, Lahore. Participants who meet the inclusion criteria will be enrolled and allocated in group A & B through sealed envelope method by Non-probability Convenient random sampling technique. Subjects in Group A will receive Instrument Assisted Soft Tissue Mobilization. Group B will receive Therapeutic Cupping. Players will be assessed by Numeric pain rating scale, Universal Goniometer and Sit & Reach Test after the completion of treatment at 6 weeks.

The data will be analyzed by SPSS, version 25. Statistical significance is P=0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age (18-25),Male Gender Only,
* Football Players, Bilateral Hamstring Tightness,
* Previous hamstring injury in the last 6 months,
* Positive SLR test,
* Positive Passive/Active Knee Extension test

Exclusion Criteria:

* Malignancy of lower limb,
* History of Lower Limb fracture in the last 6 months,
* Post-surgical condition from past 6 months,
* Neurological Conditions such as SLE, Herpes zoster, parkinsonism, Shingles disease, Musculoskeletal disorders like adductor tendinopathy, low back pain, knee injuries, hip injuries,
* Skin Allergies.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participant should be a male football player.
Enrollment: 30 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
Hamstring pain | pre and 6 weeks post interventional
  Patient level of pain will be assessed by using Numerical Rating Scale (NRS) ranging from 0 to 10
Range of motion | pre and 6 weeks post interventional
  A goniometer is an instrument that measures the available range of motion at a joint.
Flexibility | pre and 6 weeks post interventional
  The sit and reach test will be used to assess the flexibility of the hamstring muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Sikander Naseer, DPT, Principal Investigator — Study Principal Investigator
Locations (1):
- Pakistan sports board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bridgett R, Klose P, Duffield R, Mydock S, Lauche R. Effects of Cupping Therapy in Amateur and Professional Athletes: Systematic Review of Randomized Controlled Trials. J Altern Complement Med. 2018 Mar;24(3):208-219. doi: 10.1089/acm.2017.0191. Epub 2017 Nov 29. PMID 29185802
- [Background] Cheatham SW, Baker R, Kreiswirth E. INSTRUMENT ASSISTED SOFT-TISSUE MOBILIZATION: A COMMENTARY ON CLINICAL PRACTICE GUIDELINES FOR REHABILITATION PROFESSIONALS. Int J Sports Phys Ther. 2019 Jul;14(4):670-682. PMID 31440416
- [Background] Ikeda N, Otsuka S, Kawanishi Y, Kawakami Y. Effects of Instrument-assisted Soft Tissue Mobilization on Musculoskeletal Properties. Med Sci Sports Exerc. 2019 Oct;51(10):2166-2172. doi: 10.1249/MSS.0000000000002035. PMID 31083046
- [Background] Kim J, Sung DJ, Lee J. Therapeutic effectiveness of instrument-assisted soft tissue mobilization for soft tissue injury: mechanisms and practical application. J Exerc Rehabil. 2017 Feb 28;13(1):12-22. doi: 10.12965/jer.1732824.412. eCollection 2017 Feb. PMID 28349028
- [Background] Baker RT, Nasypany A, Seegmiller JG, Baker JG. Instrument-assisted soft tissue mobilization treatment for tissue extensibility dysfunction. International Journal of Athletic Therapy and Training. 2013 Sep 1;18(5):16-21.
- [Background] Cheatham SW, Lee M, Cain M, Baker R. The efficacy of instrument assisted soft tissue mobilization: a systematic review. J Can Chiropr Assoc. 2016 Sep;60(3):200-211. PMID 27713575
- [Background] Thomas K. Blood Flow Restriction and Other Innovations in Musculoskeletal Rehabilitation. In: Endurance Sports Medicine: A Clinical Guide. Cham: Springer International Publishing; 2023. p. 237-266
- [Background] Hartnett DA. Gua sha therapy in the management of musculoskeletal pathology: a narrative review. Phys Ther Rev. 2022;27(3):169-175.
- [Background] Warren AJ, LaCross Z, Volberding JL, O'Brien MS. ACUTE OUTCOMES OF MYOFASCIAL DECOMPRESSION (CUPPING THERAPY) COMPARED TO SELF-MYOFASCIAL RELEASE ON HAMSTRING PATHOLOGY AFTER A SINGLE TREATMENT. Int J Sports Phys Ther. 2020 Aug;15(4):579-592. PMID 33354391